CLINICAL TRIAL: NCT04583475
Title: Real-life Study of How to Intensify Treatment With Xolair (OMALIZUMAB) in Chronic Spontaneous Urticaria
Acronym: INTENXO
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_19; 2019-A02662-55 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Spontaneous Urticaria, Chronic
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study whose main objective is to estimate the frequency of patients benefiting from an intensification of AOM treatment at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient having expressed non-opposition
* Affiliation to a social protection scheme (beneficiary or entitled person)
* Decision by the investigator to initiate, independently of the study, an AOM treatment for Spontaneous Chronic Urticaria that may or may not be associated with an inducible component.

Exclusion Criteria:

* Patients < 18 years of age
* Patient who had previously received AOM treatment prior to the inclusion visit
* Patients under guardianship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with SUC, for whom the indication for AOM treatment has been selected.
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients benefiting from an intensification of OMA treatment at 3 months, | At 3 months
  defined as an increase in dose (more than 300mg) and/or a reduction in the administration interval to less than 4 weeks.

SECONDARY OUTCOMES:
Patient characteristics at initiation of OMA treatment expressed as numbers and percentage of total subjects. | at baseline
Proportion of patients benefiting from an intensification of OMA treatment | Baseline, at 6 months and at 9 months
  Percentage of patients who received an OMA dose greater than 300mg per dose and/or an administration interval of less than 4 weeks apart at 0, 6 and 9 months.
Activity of urticaria (score UCT) composite | at 3, 6 and 9 months
  * Proportion of patients (numbers and percentage of total) with Satisfactory response (UCT≥12 score)
  * Proportion of patients (numbers and percentage of total) with a complete response (UCT=16 score)
  * Proportion of patients (numbers and percentage of total) with unsatisfactory response (UCT score<12)
Proportion of patients with side effect during follow-up (number and percentage of the total patients) | at 3, 6 and 9 months
Life Quality | at 3, 6 and 9 months
  Comparison of the percentage and absolute change in DLQI score (Dermatology Life Quality Index score) versus baseline between patients who received a dose escalation and patients who received a standard dose of OMA.
  The DLQI is a dermatology-specific quality of life scale validated in the UCS. It assesses the impact of the disease on different aspects of life such as symptoms, feelings, activities of daily living, leisure, work, school and personal relationships. The total score ranges from 0 to 30 points: 0-1 = No effect of urticaria on the patient's life; between 2-5 = Mild effect of urticaria on the patient's life; between 6-10 = Moderate effect of urticaria on the patient's life; between 11-20 = Very strong effect of urticaria on the patient's life and between 21-30 = Extremely strong effect of urticaria on the patient's life.
Life Quality | at 3, 6 and 9 months
  Comparison of the percentage and absolute change in Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) score versus baseline between patients who received a dose escalation and patients who received a standard dose of OMA.
  The Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) for Chronic Urticaria Quality of Life Questionnaire is a tool specifically designed to assess the quality of life of patients with Chronic Urticaria Syndrome and its variant for angioedema (AE-QoL). It is a 23-item self-administered questionnaire that asks patients to rate how often each problem affects them on a Likert scale with several options (minimum 1: not at all; maximum 5: a lot). Higher scores indicate poorer quality of life.
The angioedema activity | at 3, 6 and 9 months
  Comparison of the percentage and absolute change in AAS28score versus baseline between patients who received a dose escalation and patients who received a standard dose of OMA.
  The AAS for angioedema activity score developed by Weller et al. consists of 5 questions to assess the severity of angioedema episodes. A severity grade increasing between 0 and 3 is assigned for each question. The final score corresponds to the sum of the scores for each day over a 28-day period (ASA28) and ranges from 0-420 (ASA28).

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Staumont-Salle, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No